CLINICAL TRIAL: NCT00591448
Title: Improvement of Pain Management in Burn Patients Using Virtual Reality in Conjunction With Standard Opioids and Sedatives
Brief Title: Study in the Use of Virtual Reality as an Adjunct to Pain Control in Burn Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: H-2006-0380
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2012-10

CONDITIONS: Burn
Keywords: Thermal injury
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Virtual Reality (Experimental): Patients with burns participate in VR during occupational therapy (OT) or physical therapy (PT) sessions ranging from 2 to 9 min in length
  Interventions: Other: Virtual Reality (VR)

INTERVENTIONS:
Other: Virtual Reality (VR) — See above

SUMMARY:
The purpose of this study is to evaluate the use of Virtual Reality (VR) technology during Physical Therapy (PT) and/or Occupational Therapy (OT) for patients with burns. Research questions: Do patients have increased joint Range of Motion (ROM) and reduced pain when using VR during PT compared to PT/OT when VR is not used? Do scores on an imaging ability scale correlate with the effects of VR when used with PT/OT? Do adults and children differ in their ability to engage in the virtual world?

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the use of virtual reality (VR) technology during Physical Therapy (PT) and/or Occupational Therapy (OT) for patients with burns. Due to the pain that many burn patients experience during PT/OT, we are searching for non-medicinal methods of decreasing their pain. The question we will address is: does VR use during PT/OT help to increase Range of Motion (ROM) and decrease pain intensity?

Recovery from a trauma can be hindered by the presence of acute pain. Unfortunately for burn victims, physical and occupational therapies remains an area of significant evoked pain. PT/OT is an integral part of the burn recovery and starts early in the course of treatment. PT/OT is necessary to maintain elasticity of healing skin and thereby promote functional range of motion of affected joints. If the patient is unable to participate in PT/OT due to pain, joint contractures can occur and surgical release of the contracture can become necessary.

Although pain during PT/OT can be treated with opioids, there are several drawbacks to the use of analgesics alone. Side effects, the development of opioid tolerance, and the inability of the drugs to adequately control pain are some of the disadvantages. Supplemental use of nonpharmacologic techniques, along with opioid therapy, has been found to be effective in reducing pain and anxiety. In particular, distraction has been found to be useful to minimize burn pain (Miller, 1992; Patterson, 1995). Virtual reality, due to its immersive nature that includes sight, sound, and sometimes touch, may be an even more effective method of distraction than traditional methods such as video movies or interactive video games. To explain these non-pharmacologic analgesic effects, investigators propose that the illusion of going in to the virtual world draws the patient's attention. Conscious attention is required for the experience of pain (Chapman and Nakamura, 1999; Eccleston and Crombez, 1999). The interactive nature of the immersive virtual reality make VR unusually attention grabbing, leaving less attention available to process incoming pain signals (Hoffman, Patterson and Carrougher, 2000).

In 1996, Hunter Hoffman and David Patterson co-originated new techniques using immersive virtual reality for pain control. Virtual reality is a familiar format to children and young adults, who grew up playing videogames. Like videogames, it is an environment that is stimulated by a computer. However, in virtual reality, visual experiences are presented through special stereoscopic goggles. Virtual reality simulations can include additional sensory information, such as sound through speakers and touch through cyber-gloves. Users interact with a virtual reality environment either through a keyboard, mouse, or a specially designed device. These systems are described as "fully immersive" as the user is surrounded by virtual reality stimulation. Simulated environments have been used to mimic videogames and real-world situations, such as pilot training, driver training, museum tours, and underwater expeditions. Researchers have found that immersive virtual reality distraction can reduce patient's pain rating during severe burn wound care by 30% to 50% (Hoffman, Patterson et al., 2004; Hoffman, Patterson and Carrougher, 2000). Patients receiving adjunctive VR during physical therapy reported large reductions in the amount of time spent thinking about pain, pain intensity (worst pain) and in how unpleasant they found their pain (Hoffman, Patterson, Carrougher and Sharar, 2001). In a recent fMRI brain scan study, participants reported large reductions in subjective pain when in VR compared to no VR during their scan. The controlled laboratory fMRI study further showed that VR analgesia was accompanied by large reductions in pain-related brain activity (Hoffman, Richards et al., 2004).

The proposed study will replicate and extend the work of Hoffman, Patterson and colleagues. Using similar experimental techniques, patients will serve as their own controls to evaluate the effects of the use of VR during physical therapy/occupational therapy for burn care compare to no VR during therapy during several sessions. An imagery scale will be completed by subjects prior to the first session to determine if there is a correlation between imagery scores and the effects of the VR. This may help identify patients who will benefit from VR in the future.

Prior research has shown that some patients respond better than others to adjunct therapy than others. Caregivers may be reluctant to initiate such therapies unless they are certain it will be beneficial. Kwekkeboom has developed and tested the Imaging Ability Questionnaire (IAQ) and the Kids Imaging Ability Questionnaire (KIAQ) to help determine who would benefit from this type of intervention (Kwekkeboom, Maddox, West, 2000). Participants will be completing these questionnaires prior to the first VR therapy session. The instruments for both groups will be the same with the exception of the "imaging ability". Each group will complete an "imaging ability", but one has been designed especially for children, the other for adults.

The majority of the research using VR has been focused on children. Children and adolescents are accustom to playing video games and may have an easier transition into the VR world. We are interested in the adult's ability to become engaged in VR compared to children.

Potential benefits include:

Speedier Physical Rehabilitation a Decreased Pain Experience During Necessary Care Decreased Pain Med Requirements Addition of Variety to Daily Activities Altruistic Benefit Derived From the Possible Future Benefit to Others.

ELIGIBILITY:
Inclusion Criteria:

* Able to complete subjective evaluations of pain
* English-speaking
* Not demonstrating delirium, psychosis, or any form of Organic Brain Disorder
* Able to communicate orally
* Pain associated with PT/OT
* Age six years and above

Exclusion Criteria:

* Incapable of indicating subjective evaluation of pain
* Non-English-speaking
* Severe head or neck injury or other medical conditions that prohibit patient from wearing VR helmet.
* Demonstrating delirium, psychosis, or Organic Brain Disorder
* Unable to communicate verbally
* Significant developmental disability
* Extreme susceptibility to motion sickness
* Reports having no pain/full range of motion during physical therapy
* Seizure disorder
* Frostbite

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-10; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Improved pain scores | 18 months

SECONDARY OUTCOMES:
There are no secondary outcomes | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Lee Faucher, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- United States, Madison, Wisconsin, United States